CLINICAL TRIAL: NCT00436202
Title: Evaluation of an Intervention Program for the Prevention of Anemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wolfson Medical Center (Other Government)
Collaborators: Tel Aviv District of the Health Office (Unknown)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Anemia
Record Dates: First submitted 2007-02-15; First posted 2007-02-16 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Anemia
Keywords: Anemia; Iron; Supplement
MeSH Terms: conditions — Anemia | interventions — Iron-Dextran Complex

INTERVENTIONS:
Behavioral: Iron supplement

SUMMARY:
The purpose of the study is to determine whether improvement in the accessibility to iron supplement will decrease anemia rates in infants.

DETAILED DESCRIPTION:
Iron deficiency anemia is the most common type of anemia in infants, children and women of reproductive age. The most frequent cause of iron deficiency in infants at 6 months of life is poor nutrition during a period of rapid growth and a diet lacking in iron rich foods. Children who suffered from anemia in infancy demonstrated slower cognitive development, were low achievers in school and had a high rate of behavioral disturbances.

The Ministry of Health implements a primary prevention program for anemia. If by making iron supplements more accessible would increase parental compliance in acquisition of the iron supplement and subsequently reduce the rate of iron deficiency anemia, the result would be the immediate application of the finding. It is possible to implement a program whereby the supplement will be directly available at the family health centers for purchase by the parent.

ELIGIBILITY:
Inclusion Criteria:

* Infant who visit Family Health Centers

Min Age: 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Tamar Shohat, M.D., MPH, Principal Investigator — Tel Aviv District of the Health Office
Locations (1):
- Tel Aviv District of the Health Office, Tel Aviv, Israel